CLINICAL TRIAL: NCT07294612
Title: Use of Platelet-Rich Fibrin in Bladder Exstrophy Repair: A Prospective Study
Brief Title: Use of Platelet-Rich Fibrin in Bladder Exstrophy Repair
Acronym: PRF-BEEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Medical Center, Uzbekistan (Other)
Responsible Party: Principal Investigator, Zafar Abdullaev, Head of Pediatric urology department, National Children's Medical Center, Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: №:052022/14
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Bladder Exstrophy-Epispadias Complex
Keywords: Platelet-Rich Fibrin; Bladder Exstrophy; Penopubic Fistula; Pediatric Urology; Randomized Controlled Trial; Wound Healing
MeSH Terms: conditions — Bladder Exstrophy and Epispadias Complex; Bladder Exstrophy

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled trial in which participants were assigned in a 1:1 ratio to either receive autologous platelet-rich fibrin during bladder exstrophy repair or undergo standard surgical closure without PRF. Outcomes were compared between the two independent groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Group (Experimental): Participants undergo primary bladder exstrophy repair with intraoperative application of autologous platelet-rich fibrin over the bladder neck before pubic symphysis closure.
  Interventions: Biological: Autologous Platelet-Rich Fibrin
- Non-PRF Group (Active Comparator): Participants undergo standard primary bladder exstrophy repair without the use of platelet-rich fibrin.
  Interventions: Procedure: Standard Surgical Closure

INTERVENTIONS:
Biological: Autologous Platelet-Rich Fibrin — Autologous platelet-rich fibrin prepared intraoperatively from 5-10 mL of the patient's venous blood using centrifugation at (3000 rpm for 10 min) to produce a PRF and applied over the bladder neck before pubic symphysis closure during primary bladder exstrophy repair.
  Arms: PRF Group
Procedure: Standard Surgical Closure — Standard primary bladder exstrophy repair closure performed without the use of platelet-rich fibrin.
  Arms: Non-PRF Group

SUMMARY:
Bladder exstrophy-epispadias complex (BEEC) is a rare condition in which the bladder and surrounding structures do not form normally. Surgery is required to close the bladder and restore normal anatomy, but complications such as penopubic fistula and wound breakdown are common after repair. Platelet-rich fibrin (PRF) is a material obtained from a patient's own blood that contains healing factors and may improve wound healing.

This prospective randomized controlled study evaluates whether applying autologous PRF during primary bladder exstrophy repair can reduce postoperative complications compared with standard surgical closure alone. Twenty pediatric patients with primary BEEC undergoing surgical repair were randomly assigned to either a PRF group or a non-PRF (control) group. The main outcome measured was the occurrence of penopubic fistula after surgery, along with other postoperative complications. The results of this study aim to help determine whether PRF is a safe and effective adjunct in bladder exstrophy repair.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized controlled clinical trial conducted in the Pediatric Urology Department of the National Children's Medical Center between 2022 and 2025. The study enrolled 20 male patients with primary bladder exstrophy-epispadias complex undergoing initial surgical repair. Patients with cloacal variants and complicated cases were excluded.

Participants were randomly allocated using a computer-generated random number sequence into two groups: the PRF group (n = 12), in which autologous platelet-rich fibrin was applied during bladder neck repair, and the non-PRF control group (n = 8), in which standard wound closure was performed without PRF.

In the PRF group, 5-10 mL of venous blood was collected intraoperatively and centrifuged to prepare a PRF membrane, which was applied over the bladder neck before pubic symphysis closure. Both groups underwent standardized surgical repair techniques, including complete primary repair or modified staged repair as indicated.

The primary outcome was the incidence of penopubic fistula formation. Secondary outcomes included wound dehiscence, hospital stay, and postoperative complications. Patients were followed postoperatively according to the institutional protocol.

This study was approved by the Institutional Review Board of the National Children's Medical Center (Approval No.: 052022/14), and informed consent was obtained from the parents or legal guardians of all participants.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with primary bladder exstrophy-epispadias complex (BEEC)
* Age from birth up to 18 years
* Patients undergoing primary surgical repair of bladder exstrophy
* Written informed consent provided by parents or legal guardians

Exclusion Criteria:

* Patients with cloacal variants of bladder exstrophy
* Patients with complicated or recurrent bladder exstrophy
* Patients who previously underwent bladder exstrophy repair
* Patients with severe associated congenital anomalies that could affect wound healing
* Patients with coagulation abnormalities
* Patients with severe anemia

Ages: 6 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Penopubic Fistula | from 3 month to 6 month
  Occurrence of clinically confirmed penopubic fistula following primary bladder exstrophy repair in the PRF and non-PRF groups.

SECONDARY OUTCOMES:
Incidence of Wound Dehiscence | Within 6 months after surgery
  Occurrence of postoperative wound dehiscence after primary bladder exstrophy repair in the PRF and non-PRF groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zafar, Tashkent, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohan Ehrenfest DM, Rasmusson L, Albrektsson T. Classification of platelet concentrates: from pure platelet-rich plasma (P-PRP) to leucocyte- and platelet-rich fibrin (L-PRF). Trends Biotechnol. 2009 Mar;27(3):158-67. doi: 10.1016/j.tibtech.2008.11.009. Epub 2009 Jan 31. PMID 19187989
- [Result] Kajbafzadeh AM, Abolghasemi H, Eshghi P, Alizadeh F, Elmi A, Shafaattalab S, Dianat S, Amirizadeh N, Mohseni MJ. Single-donor fibrin sealant for repair of urethrocutaneous fistulae following multiple hypospadias and epispadias repairs. J Pediatr Urol. 2011 Aug;7(4):422-7. doi: 10.1016/j.jpurol.2010.06.004. Epub 2010 Jul 15. PMID 20634140
- [Result] Guinot A, Arnaud A, Azzis O, Habonimana E, Jasienski S, Fremond B. Preliminary experience with the use of an autologous platelet-rich fibrin membrane for urethroplasty coverage in distal hypospadias surgery. J Pediatr Urol. 2014 Apr;10(2):300-5. doi: 10.1016/j.jpurol.2013.09.026. Epub 2013 Nov 13. PMID 24325905
- [Result] Soyer T, Cakmak M, Aslan MK, Senyucel MF, Kisa U. Use of autologous platelet rich fibrin in urethracutaneous fistula repair: preliminary report. Int Wound J. 2013 Jun;10(3):345-7. doi: 10.1111/j.1742-481X.2012.00983.x. Epub 2012 May 9. PMID 22568526